CLINICAL TRIAL: NCT02974543
Title: Combined Auditory-Somatosensory Stimulation to Alleviate Tinnitus
Brief Title: Auditory-somatosensory Stimulation to Alleviate Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Wallace H Coulter Center for Translational Research (Other)
Responsible Party: Principal Investigator, Susan E. Shore, Professor, Otolaryngology, Molecular and Integrative Physiology; Professor, Biomedical Engineering Kresge Hearing Research Institute The Joseph Hawkins Collegiate Research Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM00088432
Record Dates: First submitted 2016-11-14; First posted 2016-11-28 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Tinnitus
Keywords: tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham 1st (Auditory only) then Active (Bimodal) (Other): To mitigate potential placebo effects, subjects receive both a sham treatment and an active treatment. The subjects will be blinded to which treatment they are receiving. Both treatments are delivered using a take-home device programmed in the lab.
  During active treatment, the device will deliver electric somatosensory and auditory stimulation.
  Interventions: Device: Sham Treatment: unimodal auditory stimulation; Device: Active Treatment: Bimodal auditory-somatosensory stimulation
- Active (Bimodal) then Sham (Auditory only) (Other): During active treatment, the device will deliver electric somatosensory and auditory stimulation.
  To mitigate potential placebo effects, subjects receive both a sham treatment and an active treatment. The subjects will be blinded to which treatment they are receiving. Both treatments are delivered using a take-home device programmed in the lab.
  Interventions: Device: Sham Treatment: unimodal auditory stimulation; Device: Active Treatment: Bimodal auditory-somatosensory stimulation

INTERVENTIONS:
Device: Sham Treatment: unimodal auditory stimulation — All subjects will be told they will receive either Sham or Active Treatment, but will not know which treatment is assigned. Set up for the sham treatment is the same as the active treatment.
Device: Active Treatment: Bimodal auditory-somatosensory stimulation — Somatosensory stimulation will be delivered by pads positioned on the cheek overlying the trigeminal ganglion, the juncture of the temporomandibular joint or on the neck at overlying cervical nerves, c1 or c2, determined by the manner in which the subject can modulate the tinnitus.
  The auditory stimulus will be individualized based on subject baseline audiogram and tinnitus test results and is presented through a calibrated earphone.

SUMMARY:
The purpose of this study is to develop and test a subject operated device to lessen tinnitus (ringing in the ear), based on subject-feedback for stimulus presentation.

DETAILED DESCRIPTION:
This study consented 35 adult subjects. 21 subjects qualified and were randomized into the study. This project will develop and test a device with the ultimate goal of providing a patient operated device to alleviate phantom sound perception, or tinnitus, based on patient-feedback for stimulus presentation.

The device, an electrical-acoustical stimulus timing, is based on physiological findings of stimulus-timing-dependent plasticity in somatosensory and auditory nuclei,that when aberrant, contribute to tinnitus.

ELIGIBILITY:
Inclusion Criteria:

1. Constant, subjective, preferably unilateral tinnitus without any active external or middle ear pathology.
2. Hearing thresholds better than 50dB HL at peak tinnitus frequencies.
3. Able to modulate their tinnitus with a somatic maneuver
4. BothersomeTinnitus.

Exclusion Criteria:

* No participation in a tinnitus treatment regimen within the past four weeks
* Retrocochlear pathology/ VIIIth nerve lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shore, Ph.D, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Kresge Hearing Research Institute, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 14 participants consented to the study, but were screened out of allocation to either arm for excess hearing loss, lack of somatosensory modulation, or unwillingness to participate (largely due to time committments/availability).
Groups:
- Sham 1st (Auditory Only) Then Active (Bimodal): To mitigate potential placebo effects, subjects receive both a sham treatment and an active treatment. The subjects will be blinded to which treatment they are receiving. Both treatments are delivered using a take-home device programmed in the lab.
  During active treatment, the device will deliver electric somatosensory and auditory stimulation.
  Sham Treatment: unimodal auditory stimulation: All subjects will be told they will receive either Sham or Active Treatment, but will not know which treatment is assigned. Set up for the sham treatment is the same as the active treatment.
  Active Treatment: Bimodal auditory-somatosensory stimulation: Somatosensory stimulation will be delivered by pads positioned on the cheek overlying the trigeminal ganglion, the juncture of the temporomandibular joint or on the neck at overlying cervical nerves, c1 or c2, determined by the manner in which the subject can modulate the tinnitus.
  The auditory stimulus will be individualized based on s
- Active (Bimodal) Then Sham (Auditory Only): During active treatment, the device will deliver electric somatosensory and auditory stimulation.
  To mitigate potential placebo effects, subjects receive both a sham treatment and an active treatment. The subjects will be blinded to which treatment they are receiving. Both treatments are delivered using a take-home device programmed in the lab.
  Sham Treatment: unimodal auditory stimulation: All subjects will be told they will receive either Sham or Active Treatment, but will not know which treatment is assigned. Set up for the sham treatment is the same as the active treatment.
  Active Treatment: Bimodal auditory-somatosensory stimulation: Somatosensory stimulation will be delivered by pads positioned on the cheek overlying the trigeminal ganglion, the juncture of the temporomandibular joint or on the neck at overlying cervical nerves, c1 or c2, determined by the manner in which the subject can modulate the tinnitus.
  The auditory stimulus will be individualized based on s
Period: Overall Study
Arm/Group | Sham 1st (Auditory Only) Then Active (Bimodal) | Active (Bimodal) Then Sham (Auditory Only)
Started | 11 | 10
Began Washout Period | 10 | 10
Began Crossover Assignment | 10 | 10
Completed | 10 | 10
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data are included only for those participants for whom outcome measure data was completed (N=20). One subject was consented and began the study, but withdrew after week one.
Groups:
- Active 1st (Bimodal) Then Sham (Auditory Only): During active treatment the device will deliver electric somatosensory and auditory stimulation. To mitigate potential placebo effects, subjects receive both a sham treatment and an active treatment. The subjects will be blinded to which treatment they are receiving. Both treatments are delivered using a take-home device programmed in the lab. Sham Treatment: unimodal auditory stimulation: All subjects will be told they will receive either Sham or Active Treatment, but will not know which treatment is assigned. Set up for the sham treatment is the same as the active treatment. Active Treatment: Bimodal auditory-somatosensory stimulation: Somatosensory stimulation will be delivered by pads positioned on the cheek overlying the trigeminal ganglion, the juncture of the temporomandibular joint or on the neck at overlying cervical nerves, determined by how the subject can modulate the tinnitus. The auditory stimulus will be individualized based on subjects' tinnitus spectrum.
- Sham 1st (Auditory Only) Then Active (Bimodal): To mitigate potential placebo effects, subjects receive both a sham treatment and an active treatment. The subjects will be blinded to which treatment they are receiving. Both treatments are delivered using a take-home device programmed in the lab. During active treatment, the device will deliver electric somatosensory and auditory stimulation. Sham Treatment: unimodal auditory stimulation: All subjects will be told they will receive either Sham or Active Treatment, but will not know which treatment is assigned. Set up for the sham treatment is the same as the active treatment. Active Treatment: Bimodal auditory-somatosensory stimulation: Somatosensory stimulation will be delivered by pads positioned on the cheek overlying the trigeminal ganglion, the juncture of the temporomandibular joint or on the neck at overlying cervical nerves, determined by how the subject can modulate the tinnitus. The auditory stimulus will be individualized based on subjects' tinnitus spectrum.
- Total: Total of all reporting groups
Arm/Group | Active 1st (Bimodal) Then Sham (Auditory Only) | Sham 1st (Auditory Only) Then Active (Bimodal) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Tinnitus Functional Index (TFI) [Mean (Standard Deviation); unit: units on a scale] — Baseline measure of TFI score. TFI is a clinical questionnaire that assesses tinnitus impact on a subject's quality of life. It uses a scale of 0 - 100 where 0 means no negative impact on quality of life from tinnitus and 100 is devastating impact. This measure will be performed at baseline, as well as time points following active, washout, or sham periods.
  units on a scale | 34.88 (16.70) | 26.66 (14.78) | 31.78 (16.70)
Tinnitus Loudness [Mean (Standard Deviation); unit: dB] — Tinnitus matching loudness score at baseline assessment. Subjects are guided through a self-directed computerized assessment software that estimates how loud (in decibels/dB) they perceive their tinnitus to be (TinnTester). This measure will be performed at baseline, as well as time points following active, washout, or sham periods.
  dB | 58.99 (14.77) | 49.85 (18.25) | 54.42 (14.77)

OUTCOME MEASURES:

1. Primary Outcome: Change in TFI (Tinnitus Functional Index) After Treatment or Sham Compared to Baseline
Description: Change in TFI score (mean of weekly assessments for 4 weeks) from baseline for treatment and sham groups. TFI is a clinical questionnaire that assesses tinnitus impact on a subject's quality of life. It uses a scale of 0 - 100 where 0 means no negative impact on quality of life from tinnitus and 100 is devastating impact It will be administered weekly through out the study.
Time Frame: Four weeks on treatment (or sham)
Population: First 3 columns represent the data from same 10 subjects at different time points who participated in the first arm (received active treatment before sham treatment). The last 3 columns represent data from the other 10 subjects at the same timepoints who participated in the 2nd arm (received sham treatment before active treatment).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Before Sham | Washout After Active | Sham After Active | Sham Before Active | Washout After Sham | Active After Sham
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
units on a scale | -10.08 (6.79) | -5.40 (4.11) | 0.95 (10.32) | -4.34 (4.11) | -2.24 (4.58) | -5.27 (6.46)
Statistical Analysis 1: Comparison: Active Before Sham vs Washout After Active vs Sham After Active vs Sham Before Active vs Washout After Sham vs Active After Sham; Test type: Superiority; p < 0.05, Mixed Models Analysis

2. Primary Outcome: Change in Tinnitus Loudness as Assessed by TinnTester
Description: Change in Tinnitus matching loudness score (mean of weekly assessments for 4 weeks) from baseline tinnitus matching loudness score, for treatment and sham groups. Subjects are guided through a self-directed computerized assessment software that estimates how loud (in decibels) they perceive their tinnitus to be (TinnTester). This measure was performed at baseline, as well as time points following active, washout, or sham periods.
Time Frame: 4 weeks on treatment (or sham)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Active Before Sham | Washout After Active | Sham After Active | Sham Before Active | Washout After Sham | Active After Sham
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
dB | -8.25 (9.69) | -1.52 (7.16) | -3.17 (5.02) | -3.34 (4.50) | -1.67 (3.98) | -7.85 (8.79)
Statistical Analysis 1: Comparison: Active Before Sham vs Washout After Active vs Sham After Active vs Sham Before Active vs Washout After Sham vs Active After Sham; Test type: Superiority; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 12 weeks of treatment or sham
Arm/Group | Active Before Sham | Washout After Active | Sham After Active | Sham Before Active | Washout After Sham | Active After Sham
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/11 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/11 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes